CLINICAL TRIAL: NCT03956056
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Neoantigen Peptide Vaccine Strategy in Pancreatic Cancer Patients Following Surgical Resection and Adjuvant Chemotherapy
Brief Title: Neoantigen Peptide Vaccine Strategy in Pancreatic Cancer Patients Following Surgical Resection and Adjuvant Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding/staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201908124; P50CA196510-03 (NIH)
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Cancer; Pancreatic Cancer; Cancer of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — poly ICLC; Blood Specimen Collection; Monitoring, Immunologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoantigen Peptide Vaccine (Experimental): The schedule for vaccination will be Days 1, 4, 8, 15, and 22 (delays of up to 96 hours are allowed for each dose based on the adverse events experienced). Additional vaccinations will be given on Days 50 and 78 (+/- 2 weeks). The first vaccine dose may be administered following confirmation of disease-free status and within 90 days following date of repeat imaging. All study injections will be given subcutaneously and co-administered with poly-ICLC by a trained healthcare provider.
  Interventions: Biological: Neoantigen Peptide Vaccine; Drug: Poly ICLC; Procedure: Blood for immune monitoring

INTERVENTIONS:
Biological: Neoantigen Peptide Vaccine — • Each pool of vaccine study drug + poly IC:LC will be administered to one of the four limbs (A - Right Arm, B - Left Arm, C - Right Leg, D - Left Leg) by subcutaneous (SC) injection.
Drug: Poly ICLC — • Each pool of vaccine study drug + poly IC:LC will be administered to one of the four limbs (A - Right Arm, B - Left Arm, C - Right Leg, D - Left Leg) by subcutaneous (SC) injection.
  Other Names: Poly-ICLC; Hiltonol
Procedure: Blood for immune monitoring — -Baseline, day 1, day 22, day 50, day 78, week 25, and week 73

SUMMARY:
This is a phase 1 open-label study to evaluate the safety and immunogenicity of a neoantigen peptide vaccine strategy in pancreatic cancer patients following surgical resection and adjuvant chemotherapy. The neoantigen peptide vaccines will incorporate prioritized neoantigens and personalized mesothelin epitopes and will be co-administered with poly-ICLC. The hypothesis of this study is that neoantigen peptide vaccines will be safe and capable of generating measurable neoantigen-specific CD4 and CD8 T cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma; mixed histology will be included as long as the predominant histology is adenocarcinoma.
* Completed an R0 or R1 surgical resection as determined by pathology
* Pathology review demonstrates tumor cellularity no less than 30% in quantities sufficient to obtain 6-8 1mm biopsies from the original FFPE blocks.
* At least 18 years of age.
* Life expectancy of > 12 months.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * WBC>=3,000/μL
  * absolute neutrophil count>=1,500/μL
  * platelets>=100,000/μL
  * total bilirubin≤1.5 X institutional upper limit of normal (subjects with Gilbert's syndrome may be enrolled despite a total bilirubin level >1.5 mg/dL if their conjugated bilirubin is <1.5 x ULN)
  * AST≤ X institutional upper limit of normal
  * creatinine≤1.5 X institutional upper limit of normal
* International Normalized Ratio (INR) and activated partial thromboplastin time (PTT) < 1.5 x ULN provided the patient is not on anticoagulation therapy.

  9-Patients who have had a stent placed for biliary obstruction can be included in the study provided serum bilirubin at time of enrollment is within protocol limits.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Evidence of neuroendocrine tumor, duodenal adenocarcinoma, or ampullary adenocarcinoma.
* Received neoadjuvant chemotherapy for their pancreatic adenocarcinoma
* Evidence of disease recurrence or metastasis following surgical resection at any time prior to the first vaccination administration. Most patients will undergo restaging midway through adjuvant chemotherapy and at the completion of therapy; however, timing of imaging is at the discretion of the patient's medical oncologist.
* History of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only, carcinoma in situ of the cervix, or LCIS/DCIS of the breast
* Known allergy, or history of serious adverse reaction to vaccines or TLR agonists such as anaphylaxis, hives, or respiratory difficulty.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, hepatic renal, and/or other functional abnormality that would jeopardize the health and safety of the participant as determined by the investigator based on medical history, physical examination, laboratory values, and/or diagnostic studies.
* A psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator from the medical history, physical exam, and/or medical record
* Prior or currently active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication (e.g., corticosteroids) which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines. In the case of asthma or chronic obstructive pulmonary disease taking inhaled corticosteroids that does not require daily systemic corticosteroids is acceptable. Additionally, local acting steroids (topical, inhaled, or intraarticular) will be allowed. Patients on intermittent or short course steroids will be allow if the dose does not exceed 4 mg of dexamethasone (or equivalent) per day for > 7 consecutive days. Any patients receiving steroids should be discussed with the PI to determine if eligible.
* Pregnant and/or breastfeeding.
* Known HIV-positive status. These patients are ineligible because of the potential inability to generate an immune response to vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoantigen Peptide Vaccine
Started | 12
Completed | 9
Not Completed | 3
Not completed — Cannot make vaccine due to lack of tissue variants | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoantigen Peptide Vaccine
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety of Neoantigen Peptide Vaccine as Measured by the Number of Serious Adverse Events
Description: -Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0.
Time Frame: Through 30 days following completion of treatment (median follow-up of 107 days, full range of 88-157 days)
Population: 2 participants were not evaluable for this outcome measure as they did not start vaccine treatment.
Measure: Number; unit: participants
Arm/Group | Neoantigen Peptide Vaccine
Number analyzed (Participants) | 10
participants
  Grade 3 ascites | 1
  Grade 3 anemia | 1

2. Secondary Outcome: Number of Participants With Immune Response as Measured by ELISPOT Analysis
Description: The ELISpot assay was performed after in vitro culture of patient PBMC with neoantigen peptide for ~12 days. The number of spot-forming T cells, a surrogate for the number of neoantigen-specific T cells, was determined after neoantigen peptide re-stimulation for the duration of the assay (48 hours) and compared to that of control cells that were not re-stimulated with neoantigen during the assay. Independent t tests between pre- and post-vaccination PBMCs were performed.
Time Frame: Baseline through week 52
Population: 3 participants were not evaluable for this outcome measure. 2 participants were not enrolled but vaccine wasn't able to be made due to lack of tissue variants. 1 participant did not complete treatment due to disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoantigen Peptide Vaccine
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Number of Participants With Immune Response as Measured by Multiparametric Flow Cytometry (CD4)
Description: Multiparametric flow cytometry was performed as a second readout to characterize the neoantigen-specific T cell response. Markers included CD4, CD8, IFNγ, and a viability marker. After culture, as described above, T cells were stimulated overnight with/without neoantigen and stained with fluorescent antibodies specific for the various markers. Data were analyzed by comparing, between pre- and post-vaccination PBMCs, the percent ratio of IFNγ+ CD4/CD8 cells with neoantigen stimulation over those without stimulation; a >2-fold increase in response after vaccination was considered positive.
Time Frame: Baseline through week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Neoantigen Peptide Vaccine
Number analyzed (Participants) | 9
Participants | 5

4. Secondary Outcome: Number of Participants With Immune Response as Measured by Multiparametric Flow Cytometry (CD8)
Description: as for outcome 3
Time Frame: Baseline through week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Neoantigen Peptide Vaccine
Number analyzed (Participants) | 9
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days following the last day of treatment (approximately day 108).
Arm/Group | Neoantigen Peptide Vaccine
All-Cause Mortality (participants affected / at risk) | 4/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoantigen Peptide Vaccine (N=10)
Anemia (Blood and lymphatic system disorders) | 1
Ascites (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoantigen Peptide Vaccine (N=10)
Anemia (Blood and lymphatic system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Cataract correction surgery (Eye disorders) | 1
Belching (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Sore under tongue (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Body aches (General disorders) | 1
Chills (General disorders) | 3
Chills (intermittent) (General disorders) | 1
Edema at injection site (General disorders) | 5
Fatigue (General disorders) | 5
Fever (General disorders) | 4
Hip pain (General disorders) | 1
Injection site pain (General disorders) | 2
Injection site reaction (General disorders) | 4
Left knee pain (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain at surgical site (General disorders) | 1
Right buttock pain (General disorders) | 1
Shoulder pain (General disorders) | 1
Urine pain (General disorders) | 1
COVID-19 infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 1
White blood cell count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Body odor (Skin and subcutaneous tissue disorders) | 1
Bruising at injection site (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash on arms (Skin and subcutaneous tissue disorders) | 1
Skin rash on hands (Skin and subcutaneous tissue disorders) | 1
Skin redness on injection sites (Skin and subcutaneous tissue disorders) | 5
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 5
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT03956056/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03956056/ICF_001.pdf